CLINICAL TRIAL: NCT02863458
Title: Effectiveness of DNA Hypomethylating Agents and Lenalidomide in Elderly Patients With Myeloid Malignancies in the United States
Brief Title: DNA Hypomethylating Agents and Lenalidomide in Elderly Patients With Myeloid Malignancies in the US
Status: Withdrawn | Type: Observational
Why Stopped: Study was a data review, no patient recruitment occurred.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-1066
Record Dates: First submitted 2015-09-13; First posted 2016-08-11 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: MDS; AML; hypomethylating agents (HMA); Surveillance Epidemiology and End Results (SEER)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to comprehensively analyze data from a large and unselected older AML population in the US, both treated and untreated. These data will widen understanding of treatment decisions for the older Acute Myeloid Leukemia (AML) population. Through use of the SEER-Medicare Registry, the effectiveness and impact of HMA treatments as well as the effectiveness of lenalidomide will be studied.

DETAILED DESCRIPTION:
This will be the first study to comprehensively analyze data from a large and unselected older AML population in the US, both treated and untreated. These data will widen understanding of treatment decisions for the older AML population and shed light on the impact of HMA in this vulnerable population. The findings from this study will help identify the role of HMA (with its salient features of better tolerability and lesser toxicity) as a new treatment paradigm for older AML patients and enable comparison of outcomes with HMA vs other "conventional" leukemia therapies (intensive chemotherapy, low dose cytarabine or best supportive care). Additionally, with updated SEER-Medicare file carrying Medicare claims through 2013, this study will help analyze several long term outcome measures extending up to eight years for MDS patients treated with lenalidomide. Finally, the effectiveness of HMA in the SEER-Medicare MDS population will be studied by using SEER-Medicare data. This registry includes information on Medicare MDS beneficiaries - a population age cohort that has the highest incidence rates for MDS and a large sample size with absolute MDS cases approaching 40000, making it the largest MDS registry in the world.

The overall sample will include cases of MDS and AML newly diagnosed between 2001 and 2011 with claims from 2000 to 2012. Investigators estimate this will include approximately 50,000 patients.Therefore, the Target Follow Up design looks at patient records over a span of 12 years. Consists of patients with myeloid malignancies diagnosed during 2001-2011 at the age of 66 years or older and alive in September 2004 (i.e. 3 months after FDA approval of azacitidine for MDS), with known month of diagnosis, and not identified from death certificates or autopsy only, who had continuous Medicare Part A and B coverage, and were not enrolled in a health maintenance organization during the period of interest. The overall sample will include cases of MDS and AML newly diagnosed between 2001 and 2011 with claims from 2000 to 2012.

Variables of interest to be collected will include: MDS subtypes, age at diagnosis, sex, race, comorbidities, median household income at the zip code level, treatments (including supportive care) from diagnosis to AML progression, transfusion status, NCI comorbidity index score, response to treatments (using International Working Group criteria), physician characteristics (speciality data),and hospital characteristics (bed size, teaching status, case volume).

ELIGIBILITY:
Inclusion Criteria:

* patients with myeloid malignancies diagnosed during 2001-2011 at the age of 66 years or older
* alive in September 2004 (i.e. 3 months after FDA approval of azacitidine for MDS)
* known month of diagnosis, and not identified from death certificates or autopsy only
* continuous Medicare Part A and B coverage, and were not enrolled in a health maintenance organization during the period of interest

Exclusion Criteria:

* Anyone under 66 years

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The overall sample will include cases of MDS and AML newly diagnosed between 2001 and 2011 with claims from 2000 to 2012. Investigators estimate this will include approximately 50,000 patients. To allow adequate time for HMA usage to begin to stabilize, our analysis will be restricted to patients alive at least 3 months after its approval. Decitabine received FDA approval for all subtypes of MDS in June 2006, but it was not covered by Medicare initially, so our analysis of it will be restricted to patients who were alive in January 2007. Patients will be followed from the date of their first MDS claim (index date) through death or study end, whichever occurred first.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants on hypomethylating agents (HMA) and the effectiveness of HMA in the SEER-Medicare MDS population | Analaysis restricted to patients alive at least 3 months after HMA approval. Patients will be followed from date of their first MDS claim (index date) through death or study end, whichever occurred first.
  Study patterns & determinants of HMA use in SEER-Medicare MDS population: Use of "2+BCBM" to ID registered & unregistered MDS cases. Map out geographical distribution of HMA use based on MDS patients reclassified by SMMRS, which will yield the proportion of higher-risk (HR) & lower-risk (LR) patients receiving HMA. Survival times to be analyzed using Cox models with time varying covariates. Predictors to be selected for both types of responses using learning interactions via hierarchical group-lasso regularization & monotone spline transformations. Utilization of non-parametric random Forest & random Survival Forest methods to build regression models & assess goodness of fit & functional form of the model-based results. Conduction of propensity score analyses of treatment effects as an alternative method for treatment-assignment bias correction. Propensity scores to be calculated using a generalized boosting method as implemented in the R package twang. Computations will be done in R.
Develop predictive models of HMA treatment outcomes using SEER-Medicare data | Analaysis restricted to patients alive at least 3 months after HMA approval. Patients will be followed from date of their first MDS claim (index date) through death or study end, whichever occurred first.
  To develop predictive models of HMA treatment outcomes using SEER-Medicare data: Treatment response analysis will include variables that are extractable from SEER-Medicare files that can be used to infer standard clinical response criteria. The outcome measures will include: 1) the proportion of patients completing an HMA therapeutic-length treatment episode (TTE) [6 cycles = ~6 months]; 2) changes in transfusion dependence; 3) the number of acute hospitalizations during the HMA therapy period; 4) the time from treatment initiation for MDS to progression to AML; and 5) overall survival from the time of HMA initiation.

SECONDARY OUTCOMES:
Effectiveness of lenalidomide in the SEER-Medicare MDS population | Analaysis restricted to patients alive at least 3 months after HMA approval. Patients will be followed from date of their first MDS claim (index date) through death or study end, whichever occurred first.
  An adequate sample size is used to undertake assessment of several variables that affect use of lenalidomide as well as treatment outcomes which aim to analyze (a) prescribing patters of lenalidomide among the low risk (LR)and high risk (HR) MDS with time (from 2006 to 2013) and consistency with clinical guidelines (b) trends in combination therapy (lenalidomide + other MDS therapies) with time (c) determinants of response to lenalidomide - underlying comorbidities, duration of treatment exposure (in terms of number of cycles), concomitant use of azacitidine or other MDS therapies with transfusion status (e) associations between lenalidomide and a variety of outcomes, including survival, progression to AML, secondary solid tumor malignancies and thromboembolic events and (e) differences in lenalidomide use and outcome between MDS Centers of Excellence (using data from MDS Clinical Consortium) versus community setting.
Identify the role of HMA (with its salient features of better tolerability and lesser toxicity) as a new treatment paradigm for older AML patients and enable comparison of outcomes with HMA vs other "conventional" leukemia therapies. | Analaysis restricted to patients alive at least 3 months after HMA approval. Patients will be followed from date of their first MDS claim (index date) through death or study end, whichever occurred first.
  To develop predictive models of HMA treatment outcomes using SEER-Medicare data: Treatment response analysis will include variables that are extractable from SEER-Medicare files that can be used to infer standard clinical response criteria. The outcome measures will include: 1) the proportion of patients completing an HMA therapeutic-length treatment episode (TTE) [6 cycles = ~6 months]; 2) changes in transfusion dependence; 3) the number of acute hospitalizations during the HMA therapy period; 4) the time from treatment initiation for MDS to progression to AML; and 5) overall survival from the time of HMA initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, MPh, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
share study data with Celgene and will plan to publish a manuscript upon completion of the study